CLINICAL TRIAL: NCT00173173
Title: Epidemiological Studies of Eating Disorders in Gifted Dance Students and Ordinary High School Students:Prevalence Rate, Risk Factors and 1-Year Outcome (1st Year).
Brief Title: Epidemiological Studies of Eating Disorders in Gifted Dance Students(1st Year)
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Other Study IDs: 9461700424; NSC-92-2314-B-002-293; NSC-91-2413-H-134-021
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2005-09-15 (Estimated); Status verified 2003-08

CONDITIONS: Eating Disorders
Keywords: Gifted dance students; eating disorders; prevalence; risk factors; BITE
MeSH Terms: conditions — Feeding and Eating Disorders; Bites and Stings

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
This is the first-year part of a two-phase prospective study. The aims of the study are to investigate the prevalence rate of eating disorders in Taiwan, it's correlated psychosocial risk factors and establish the validity index of BITE. The study subjects consist of Taiwanese gifted dance high school students and age, sex, school-matched ordinary class students. All students completed questionnaires(Eating Altitude Test(EAT-26), Bulimic Investigatory Test, Ediburgh (BITE), Body Shape Questionnaire (BSQ), Physical Appearance Related Teasing Scale, Pubertal Develoment Scale, and Brief Symptom Rating Scale (BSRS) at first phase. All subjects who are above threshold (EAT-26 score≧20 and BMI≦17.5m2; the symptom scale score of BITE≧15 and/or severity scale≧5),and 10% of the sub-threshold cases need to receive second-phase interview by two senior psychiatrists. The contents of interview included SCID-IP, and risk factors assessment for eating disorders. The known risk factors included both personal factors (history of obesity, psychiatric, menstruation, teasing, or sexual or physical abuse, etc.) as well as family factors (parental problems, history of obesity, dieting, psychiatric illness etc.).

Statistical analyses were conducted using SPSS 10.0 for Windows/PC. Categorical data were analyzed by nonparametric test (Chi-square test). ANOVA or Student's t-test was used for continuous data analyses. Reliability is assessed by internal consistency and test-retest reliability. Inter-rater reliability was assessed by Kappa statistics. The sensitivity and specificity for eating disorders were calculated for individual screening instrument.ROC analyses were undertaken to evaluate the overall performance of the BITE +/- EAT in detecting eating disorder cases. Regression analysis was applied to determine predictors of disordered eating or eating disorder status. A value of P< 0.05 was considered statistically significant.

DETAILED DESCRIPTION:
This is the first-year part of a two-phase prospective study. The aims of this study are to investigate the prevalence rate of eating disorders in Taiwan, it's correlated psychosocial risk factors and establish the validity index of BITE. The study subjects consist of Taiwanese gifted dance high school students and comparable ordinary class students. Parental informed consent for nonpartipation was delivered 3 days before study started.All students completed questionnaires(Eating Altitude Test (EAT-26), Bulimic Investigatory Test, Ediburgh (BITE), Body Shape Questionnaire (BSQ), Physical Appearance Related Teasing Scale, Pubertal Develoment Scale, and Brief Symptom Rating Scale (BSRS) at first phase. All subjects who are above threshold (EAT-26 score≧20 and BMI≦17.5Kg/m2; the symptom scale score of BITE≧15 and/or severity scale≧5),and 10% of the sub-threshold cases need to receive second-phase interview by two senior psychiatrists. The contents of interview included SCID-IP, and risk factors assessment for eating disorders. The known risk factors included both personal factors (history of obesity, psychiatric, menstruation, teasing, or sexual or physical abuse, etc.) as well as family factors (parental problems, history of obesity, dieting, psychiatric illness etc.).

Statistical analyses were conducted using SPSS 10.0 for Windows/PC. Categorical data were analyzed by nonparametric test (Chi-square test). ANOVA or Student's t-test was used for continuous data analyses. Reliability is assessed by internal consistency and test-retest reliability. Inter-rater reliability was assessed by Kappa statistics. The sensitivity and specificity for eating disorders were calculated for individual screening instrument.ROC analyses were undertaken to evaluate the overall performance of the BITE +/- EAT in detecting eating disorder cases. Regression analysis was applied to determine predictors of disordered eating or eating disorder status. A value of P< 0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* gifted dance students and ordinary high school students .

Exclusion Criteria:

-

Ages: 16 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 2200
Dates: Start 2003-08; Study Completion 2004-07

CONTACTS AND LOCATIONS:
Overall Officials: Mei-Chih Tseng, MD, Principal Investigator — National Taiwan Univetsity Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan